CLINICAL TRIAL: NCT07391826
Title: A Prospective, Randomized, Controlled, Phase II Clinical Study of Megestrol Acetate Oral Suspension for Cachexia in Patients With cStage III Gastric/Gastroesophageal Junction Adenocarcinoma Receiving Neoadjuvant Therapy With Serplulimab Combined With SOX
Brief Title: Megestrol Acetate Oral Suspension for Cachexia in Patients With cStage III Gastric/Gastroesophageal Junction Adenocarcinoma Receiving Neoadjuvant Therapy With Serplulimab Combined With SOX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEGACACHE
Record Dates: First submitted 2025-07-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-06

CONDITIONS: Stage III Gastric Cancer
Keywords: gastric/gastroesophageal junction adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): megestrol acetate oral suspension + serplulimab + SOX
  Interventions: Drug: megestrol acetate oral suspension + serplulimab + SOX
- control group (Experimental): serplulimab + SOX
  Interventions: Drug: serplulimab + SOX

INTERVENTIONS:
Drug: megestrol acetate oral suspension + serplulimab + SOX — megestrol acetate oral suspension + serplulimab + SOX
  Arms: Treatment group
Drug: serplulimab + SOX — serplulimab + SOX
  Arms: control group

SUMMARY:
This study is an open-label, prospective, randomized controlled phase II clinical study. The purpose is to evaluate the efficacy and safety of megestrol acetate oral suspension for patients with cachexia and cStage III gastric/gastroesophageal junction adenocarcinoma who receive neoadjuvant therapy with serplulimab combined with SOX. This study intends to include 48 patients with locally advanced gastric adenocarcinoma who have not received any treatment, meet the diagnosis of cachexia, and are operable as research subjects. It is expected that 32 patients will be included in the experimental group and 16 patients will be included in the control group, with an inter-group ratio of approximately 2:1. After signing the informed consent, the patients will be screened and meet the inclusion and exclusion criteria. The groups will be assigned according to the random results. The patients will receive or not receive megestrol acetate oral suspension during the 3 cycles of serplulimab SOX regimen before surgery. After the second and third cycles of medication, the efficacy of neoadjuvant therapy and the possibility of radical gastric cancer D2 resection will be evaluated by imaging examinations, and radical gastric cancer surgery will be performed within 2-6 weeks after the third dose is completed. The treatment of postoperative patients will be decided by clinicians and patients based on actual clinical diagnosis and treatment.

Patients must be given study drug treatment within 7 days after randomization. The dosing window for each cycle after the first dose is ±7 days. Before each dose, patients must complete the corresponding examinations specified in the protocol to assess the safety and tolerability of the treatment.

Dosage regimen:

* Treatment group: megestrol acetate oral suspension + serplulimab + SOX
* Control group: serplulimab + SOX

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of written informed consent;
2. Age at enrollment ≥ 18 years and ≤ 80 years;
3. Eastern Cooperative Oncology Group (ECOG, see Appendix 4) physical status score of 0-2;
4. Expected survival ≥ 6 months;
5. According to the 8th edition of AJCC gastric cancer staging, patients with cStage III (cT3-4aN1-3M0) assessed by abdominal CT and diagnosed with G/GEJ adenocarcinoma by gastroscopy and pathology, and only Siewert III type and Siewert II type subjects who do not require combined thoracotomy are allowed to be enrolled in gastroesophageal junction (GEJ) cancer;
6. Meet the diagnostic criteria for cachexia (based on Fearon diagnostic criteria).

   Diagnostic criteria for cachexia: any of the following combined with anorexia or systemic inflammatory response: (1) involuntary weight loss of >5% in 6 months; (2) BMI <18.5 kg/m2, and involuntary weight loss of >2% in 6 months; (3) limb skeletal muscle index meets the diagnostic criteria for sarcopenia (male <7.26 kg/m²; female <5.45 kg/m²), and involuntary weight loss of >2% in 6 months.
7. Before enrollment, a gastrointestinal surgeon and an imaging physician jointly evaluated and determined that the tumor was cStage III and eligible for R0 resection with the purpose of cure. The patient agreed to undergo radical surgery and was judged by the surgeon to have no contraindications to surgery;
8. No previous systemic treatment for the current disease, including surgical treatment, anti-tumor chemoradiotherapy/immunotherapy, etc.;
9. Good cardiac function, and resection with the purpose of cure can be performed. If clinically indicated, patients with underlying ischemic, valvular heart disease or other severe heart disease should be evaluated by a cardiologist before surgery;
10. Normal function of major organs
11. Female patients must meet the following requirements:

    * Menopausal (defined as no menstruation for at least 1 year, and no other confirmed cause other than menopause), or surgical sterilization (ovarian and/or uterine removal), or patients of childbearing potential must meet the following requirements at the same time:
    * A negative pregnancy test within 7 days before the first medication;
    * Agree to use contraceptive measures with an annual failure rate of < 1% or maintain abstinence (avoid heterosexual intercourse) (from signing the informed consent form to at least 120 days after the last dose of the trial drug, and at least 9 months after surgery (contraceptive methods with an annual failure rate of < 1% include bilateral tubal ligation, male sterilization, correct use of hormonal contraceptives that can inhibit ovulation, hormone-releasing intrauterine devices, and copper-containing intrauterine devices.);
    * No breastfeeding.
12. Male patients must meet the following requirements: agree to abstinence (avoid heterosexual intercourse) or take contraceptive measures. The contraceptive measures are as follows: When the partner is a woman of childbearing age or the partner is pregnant, the male patient must abstain from sex or use condoms correctly for contraception for at least 120 days after the last dose of the trial drug and at least 9 months after surgery. The reliability of sexual abstinence should be evaluated with reference to the duration of the clinical study, patient preferences, and daily lifestyle. Regular abstinence (e.g., calendar day, ovulation period, basal body temperature, or post-ovulation contraceptive methods) and ejaculation outside the body are unqualified contraceptive methods;
13. The subject read and fully understood the patient instructions and signed the informed consent form.

Exclusion Criteria:

1. The patient has had other malignant tumors in the past (within 5 years) or concurrently. Patients with cured localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, stage I lung cancer, stage I colorectal cancer, etc. can be included in the group;
2. Patients who are preparing for or have received organ or bone marrow transplantation in the past;
3. Patients who have received blood transfusion within 2 weeks before the first medication, or have a history of bleeding, and have any severe bleeding events of grade 3 or above in CTCAE5.0 within 4 weeks before screening;
4. Patients with abnormal coagulation function and bleeding tendency (INR is in the normal value > 1.5 without the use of anticoagulants); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogs; On the premise that the international normalized ratio (INR) of prothrombin time is ≤1.5, low-dose warfarin (1 mg orally, once a day) or low-dose aspirin (daily dose not exceeding 100 mg) is allowed for preventive purposes;
5. Arterial/venous thrombotic events within 6 months before screening, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis (except for venous thrombosis caused by intravenous catheterization during previous chemotherapy, which is judged by the researcher to have been cured) and pulmonary embolism;
6. Myocardial infarction and poorly controlled arrhythmia (including QTc interval ≥450 ms for men and ≥470 ms for women) within 6 months before the first medication (QTc interval is calculated by Fridericia formula);
7. NYHA standard III-IV heart failure or cardiac ultrasound examination: LVEF (left ventricular ejection fraction) <50%;
8. Urinalysis indicates urine protein ≥++ and confirms that the 24-hour urine protein quantification is >1.0 g;
9. Pleural effusion or peritoneal effusion with clinical symptoms that require clinical intervention;
10. Human immunodeficiency virus (HIV) infection;
11. Active pulmonary tuberculosis;
12. Long-term unhealed wounds or incompletely healed fractures;
13. Patients with past or current interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe lung function impairment, etc., which may interfere with the detection and treatment of suspected drug-related pulmonary toxicity;
14. Patients with known active or suspected autoimmune diseases, except those who are in a stable state of the disease at the time of enrollment (systemic immunosuppressant therapy is not required);
15. Patients with a history of severe chronic autoimmune diseases, such as systemic lupus erythematosus, etc.; patients with a history of inflammatory bowel diseases such as ulcerative colitis and Crohn's disease, and a history of chronic diarrheal diseases such as irritable bowel syndrome; patients with a history of sarcoidosis or tuberculosis; patients with a history of active hepatitis B, hepatitis C, and HIV infection; patients with well-controlled non-severe immune diseases, such as dermatitis, arthritis, psoriasis, etc. can be enrolled. Patients with hepatitis B virus titer < 500 copies/ml can be enrolled;
16. Patients who need to receive systemic corticosteroids (> 10 mg/day prednisone effective dose) or other immunosuppressive drugs within 14 days before the first medication or during the study. However, the following conditions are allowed to be enrolled: In the absence of active autoimmune diseases, patients are allowed to use topical or inhaled steroids, or adrenal hormone replacement therapy with a dose of ≤ 10mg/day prednisone effective dose;
17. Any active infection requiring systemic anti-infective treatment within 14 days before the first medication, except for prophylactic antibiotic treatment (such as prevention of urinary tract infection or chronic obstructive pulmonary disease);
18. Live vaccine treatment within 28 days before the first medication, except for inactivated viral vaccine for seasonal influenza;
19. Previously received antibody/drug treatment for immune checkpoints, such as PD-1, PD-L1, CTLA-4 inhibitors, etc.;
20. Receiving other drug-related clinical research treatment; patients who are undergoing other testing or surgical clinical research can be enrolled;
21. Known history of allergy or intolerance to any study drug or its components;
22. Patients have a history of alcoholism, drug abuse and drug abuse. Patients who have stopped drinking can be included in the group;
23. Patients who do not follow the doctor's advice, do not use the medicine according to the regulations, or have incomplete information, which may affect the judgment of efficacy or safety;
24. Pregnant or lactating female patients;
25. Any condition that affects gastrointestinal absorption, such as dysphagia, a history of gastrectomy or uncontrollable vomiting; tube feeding or parenteral nutrition; anorexia nervosa, anorexia caused by mental illness or pain that makes it difficult to eat.
26. Taking or planning to take other appetite or weight-increasing drugs, such as: adrenal corticosteroids (except for short-term use of dexamethasone during chemotherapy), androgens, progesterone drugs, thalidomide, olanzapine and anamorelin or other appetite stimulants.
27. Patients with Cushing's syndrome, adrenal or pituitary insufficiency; patients with uncontrolled diabetes.
28. Postmenopausal women with a history of abnormal vaginal bleeding within one year; premenopausal women with a history of endometrial thickening (>15mm) within one year.
29. Any arterial thromboembolic event within 6 months before the first dose, venous thromboembolic event of NCI CTCAE 5.0 grade 3 or above (requiring urgent medical intervention, such as pulmonary embolism or intracardiac embolism), transient ischemic attack, cerebrovascular accident, hypertensive crisis or hypertensive encephalopathy; acute exacerbation of chronic obstructive pulmonary disease within 1 month before the first dose; current hypertension and systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg after oral antihypertensive drug treatment.
30. History of severe bleeding tendency or coagulation disorder; clinically significant bleeding symptoms within 1 month before the first dose, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing up or coughing up ≥1 teaspoon of fresh blood or small blood clots or only coughing up blood without sputum, blood in sputum is allowed), nasal bleeding (excluding epistaxis and retractile blood in nose).
31. Patients with other severe, acute and chronic diseases that may increase the risk of participating in the study and taking the study drugs, and who are judged by the researchers to be unsuitable for participating in the clinical study.
32. Other conditions that the researchers judge to be unsuitable for this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients whose weight did not decrease | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  The proportion of subjects with a weight loss of no more than 2 kg from the initiation of neoadjuvant therapy to the time immediately preceding radical surgery.

SECONDARY OUTCOMES:
appetite improve | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  The proportion of subjects whose appetite improved based on the anorexia/cachexia subscale-12，A/CS-12 scale during neoadjuvant treatment, The total score ranges from 0 to 48, with lower scores indicating poorer appetite status in patients.
Quality of life by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire(EORTC QLQ-C30) | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  The total score of this scale ranges from 0 to 100. The higher the score of the functional scale or the overall quality of life, the better the function or overall quality of life.
CRP indicators | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  The level of change in CRP during neoadjuvant treatment.
IL-6 indicators | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  The level of change in IL-6 during neoadjuvant treatment.
TNF-α indicators | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  The level of change in TNF-α during neoadjuvant treatment.
serum nutritional indicators (albumin, hemoglobin) | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  The level of change in nutritional indicators (albumin, hemoglobin) during neoadjuvant treatment.
The level of change in L3 skeletal muscle index (L3 SMI) | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  The level of change in L3 skeletal muscle index (L3 SMI) during neoadjuvant treatment.
The number of completed neoadjuvant treatment cycles | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  Three cycles of neoadjuvant therapy are planned, with assessment of whether the number of cycles is reduced due to reasons such as subject intolerance.
The number of the occurrence of drug dose reduction | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  A drug dosage reduction of more than 15% is defined as a dosage reduction.
pathological response | Assessment shall be completed within one week following radical surgery.
  Pathological complete remission (pCR) rate：It is defined as the absence of grossly visible tumor residue in gastric cancer resection specimens following neoadjuvant therapy, with no tumor cells identified microscopically after extensive sampling of the primary tumor site.

OTHER OUTCOMES:
Immune microenvironment alterations during treatment | From the date of the first neoadjuvant therapy until the date of radical surgery,assessed up to 6 months
  Assessment of the immune microenvironment is performed based on the proportions of T cell subsets.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical Unviersity, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol